CLINICAL TRIAL: NCT04123665
Title: A Clinical Study Investigating the Gingivitis Efficacy of a Test Dentifrice
Brief Title: A Phase 3 Clinical Study Investigating the Gingivitis Efficacy of a Test Dentifrice Containing Stannous Fluoride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202687
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Gingivitis
Keywords: Oral Health; Antiplaque; Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Test Dentifrice (Experimental): In this arm, participants will apply a full ribbon of dentifrice ( 0.454% w/w stannous fluoride) to the bristles of a study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) and record on their study diary completed brushings.
  Interventions: Drug: Stannous fluoride
- Control Dentifrice (Placebo Comparator): In this arm, participants will apply a full ribbon of negative control dentifrice (1000 ppm fluoride as sodium monofluorophosphate [SMFP] to the bristles of a study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) and record on their study diary completed brushings.
  Interventions: Drug: Sodium monofluorophosphate

INTERVENTIONS:
Drug: Stannous fluoride — In this arm, participants will apply a full ribbon of dentifrice ( 0.454% w/w stannous fluoride) to the bristles of a study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) and record on their study diary completed brushings.
  Arms: Experimental Test Dentifrice
Drug: Sodium monofluorophosphate — In this arm, participants will apply a full ribbon of negative control dentifrice (1000 ppm fluoride as SMFP to the bristles of a study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) and record on their study diary completed brushings.
  Other Names: Colgate Cavity Protection®, USA marketed dentifrice
  Arms: Control Dentifrice

SUMMARY:
The purpose of this study is to evaluate and compare the gingival health of a test dentifrice (0.454% weight by weight [w/w] stannous fluoride) to a negative control dentifrice by comparing modified gingival index, bleeding index and plaque index scores.

DETAILED DESCRIPTION:
This will be a single-center, examiner-blinded, randomized, stratified, two-treatment parallel group, 24-week clinical study in healthy adult volunteers with moderate gingivitis. Eligible participants will be stratified based on gender and baseline mean whole mouth modified gingival index (MGI) score (Low: less than or equal to [<=] 2.00/High greater than [>]2.00) to ensure a balance in gingivitis across both treatment groups, and then randomized into one of two treatment groups. Treatment effect will be evaluated by comparing MGI , bleeding index and plaque index scores after 12 and 24 weeks use of a dentifrice containing 0.454% w/w stannous fluoride to a negative control dentifrice. During the 24 week treatment period, participants will apply a full ribbon of dentifrice to the head of a study toothbrush and brush their teeth in their usual manner at home for one timed minute twice daily (morning and evening) and record on their study diary completed brushings.

ELIGIBILITY:
Inclusion Criteria:

* Consent :Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.
* General Health: Good general and mental health with, in the opinion of the investigator, no clinically significant and relevant abnormalities of medical history or oral examination.
* Dental Health: A minimum of 20 natural teeth and a minimum of 40 gradable surfaces for: a) MGI, BI and PI. A scorable surface is defined as a surface that has 50% of the surface gradable. Third molars, orthodontically banded/ bonded, fully crowned or extensively restored or grossly carious teeth are not included in the tooth count; b) Moderate gingivitis present at the screening visit in the opinion of the investigator; c) Mean whole mouth MGI between 1.75 and 2.30 and mean whole mouth supra-gingival PI score 1.5 at Baseline Visit.

Exclusion Criteria:

* Pregnancy and breast-feeding: Women who are known to be pregnant or who are intending to become pregnant or women who are breast-feeding over the duration of the study.
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Tobacco Use: Current smokers or smokers who have quit within the past six months, prior to screening, or participants currently using smokeless forms of tobacco - e.g. chewing tobacco.
* Concomitant Medications - Treatments Screening (Visit 1)

  1. Currently taking antibiotics or requiring antibiotic use prior to dental prophylaxis or other dental procedures.
  2. Currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
  3. Currently taking a systemic medication which, in the opinion of the Investigator, could affect gingival condition (e.g. calcium channel blockers, or aspirin therapy).
  4. Current use of a chlorhexidine mouthwash. Baseline (Visit 2)
  5. Currently taking antibiotics or taken antibiotics in the previous 14 days or requiring antibiotic use prior to dental prophylaxis or other dental procedures.
  6. Has taken an anti-inflammatory medication which, in the opinion of the investigator, could affect gingival condition in the previous 14 days.
  7. Has taken a systemic medication which, in the opinion of the investigator, could affect gingival condition in the previous 14 days (e.g. calcium channel blockers, or aspirin therapy).
* General Dentition Exclusions

  1. Current active caries or periodontitis that may, in the opinion of the investigator, compromise the study outcomes or oral health of the participants if they participate in the study.
  2. Restorations in a poor state of repair.
  3. Partial dentures or orthodontic appliances.
  4. Teeth bleaching within 12 weeks of screening.
* Clinical Study/Experimental Medication

  1. Participation in another clinical study or receipt of an investigational drug or investigational oral care product within 30 days of the Baseline Visit.
  2. Previous participation in this study.
* Substance abuse: Recent history (within the last year) of alcohol or other substance abuse.
* Personnel:

  1. Employed by the sponsor or the study site or members of their immediate family.
  2. Employed by any dentifrice manufacturer or their immediate family.
* Other Conditions: Any condition that would impact on the safety of the participant or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2013-12-11 (Actual); Study Completion 2013-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

REFERENCES:
- [Derived] Parkinson CR, Milleman KR, Milleman JL. Gingivitis efficacy of a 0.454% w/w stannous fluoride dentifrice: a 24-week randomized controlled trial. BMC Oral Health. 2020 Mar 26;20(1):89. doi: 10.1186/s12903-020-01079-6. PMID 32216778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in United States.
Pre-assignment Details: A total of 125 participants were screened for the study. Of these, 98 participants were enrolled and allocated to a randomized treatment. 27 participants were not enrolled, of which, 19 did not meet study criteria, 3 lost to follow-up and 5 withdrew their consent.
Groups:
- Experimental Test Stannous Fluoride Dentifrice: In this arm, participants applied a full ribbon of dentifrice (0.454% weight by weight [w/w] stannous fluoride) to the bristles of a study toothbrush and brushed their teeth in their usual manner for one timed minute twice daily (morning and evening) and recorded on their study diary completed brushings for 24 weeks.
- Control Sodium Monofluorophosphate Dentifrice: In this arm, participants applied a full ribbon of negative control dentifrice (1000 parts per million [ppm] fluoride as sodium monofluorophosphate [SMFP] to the bristles of a study toothbrush and brushed their teeth in their usual manner for one timed minute twice daily (morning and evening) and recorded on their study diary completed brushings for 24 weeks.
Period: Overall Study
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Started | 50 | 48
Completed | 42 | 48
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (N=98) included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (14.55) | 38.8 (12.44) | 39.2 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 43 | 39 | 82
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Baseline Modified Gingival Index (MGI) strata [Count of Participants; unit: Participants] — Participants with mean MGI score between1.75 - 2.30, a Plaque Index (PI) score >1.5 and who met all other inclusion/ exclusion criteria were stratified based on gender and baseline MGI score (Low [less than or equal to] <=2.00 or High [more than]>2.00). PI score ranges from 0-5 and MGI score ranges from 0-4. Efficacy analysis were further performed on these participants sub-grouped in the strata with their score details mentioned in their respective outcome measure. Population: A subgroup analysis using MGI stratification based upon gender
  Participants
    Male: number analyzed (Participants) | 16 | 17 | 33
    Male: MGI less than or equal to [<=] 2.00 | 5 | 5 | 10
    Male: MGI more than [>] 2.00 | 11 | 12 | 23
    Female: number analyzed (Participants) | 34 | 31 | 65
    Female: MGI less than or equal to [<=] 2.00 | 18 | 16 | 34
    Female: MGI more than [>] 2.00 | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Evaluation and Comparison of Gingival Health Measured by Bleeding Index (BI) at 24 Weeks
Description: BI-to assess bleeding elicited on probing as a measure of gingival condition. Gingivae were air dried and examiner assessed bleeding using a probe which was gently inserted into gingival crevice to depth of approximately(app)1millimeter(mm)and run around tooth(angle of app60[degrees(deg)] to long axis of tooth), gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium. BI assessed on facial and lingual gingival surfaces of each scorable tooth(7in each arch). 3scores were recorded buccally/labially,3scores lingually/palatally. All scorable teeth in one quadrant were probed first(app30seconds[sec])before recording number of gingival units which bled. Values presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values(i.e.,0-2).BI score:0=no bleeding after30sec,1=bleeding upon probing after30sec,2=immediate bleeding observed. Lower scores indicate better results.
Time Frame: At Week 24
Population: Intent-to-treat (ITT) population [N=91] included all participants who received study treatment and had at least one post-baseline efficacy measurement. Number analyzed in this outcome measure signifies those who were evaluated.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 43 | 48
Score on scale | 0.11 (0.094) | 0.19 (0.105)
Statistical Analysis 1: Comparison: Experimental Test Stannous Fluoride Dentifrice vs Control Sodium Monofluorophosphate Dentifrice; Test type: Superiority; p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) with factors for treatment group and gender, and the baseline whole mouth mean BI and whole mouth MGI as covariates; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.11 to -0.04] — Difference is first named treatment (experimental) minus second named treatment (control)

2. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by BI at 12 Weeks
Description: BI-to assess bleeding elicited on probing as a measure of gingival condition. Gingivae were air dried and examiner assessed bleeding using a probe which was gently inserted into gingival crevice to depth of app 1 mm and run around tooth (angle of app 60 deg to long axis of tooth), gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium. BI assessed on facial and lingual gingival surfaces of each scorable tooth (7in each arch). 3 scores were recorded buccally/ labially, 3scores lingually/ palatally. All scorable teeth in one quadrant were probed first (app 30 sec) before recording number of gingival units which bled. Values presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e.,0-2). BI score:0=no bleeding after 30 sec, 1=bleeding upon probing after 30 sec,2=immediate bleeding observed. Lower scores indicate better results.
Time Frame: At Week 12
Population: ITT population [N=91] included all participants who were enrolled and randomly allocated to treatment and are analyzed in the groups to which they were randomized.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 43 | 48
Score on scale | 0.11 (0.104) | 0.23 (0.124)

3. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by BI Indices in Low MGI Subgroups (<=2.00) After 12 and 24 Weeks
Description: BI-to assess bleeding elicited on probing as measure of gingival condition.Gingivae were air dried,examiner assessed bleeding using probe gently inserted into gingival crevice to depth of app.1mm and run around tooth(at angle of app.60deg to long axis of tooth),gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium.BI assessed on facial,lingual gingival surfaces of each scorable tooth(7in each arch).3scores recorded buccally/labially and 3lingually/palatally. All scorable teeth in 1quadrant probed first(app.30sec)before recording number of gingival units which bled.Participants stratified based upon gender and baseline MGI score(Low:<=2.00,High: >2.00).Whole mouth mean of BI calculated by-taking average overall tooth sites assessed;to compare magnitude of differences in two strata.BI scoring:0=no bleeding after 30sec,1=bleeding upon probing after 30sec,2=immediate bleeding observed. Lower scores- better results.
Time Frame: At Week 12 and Week 24
Population: Analysis was performed on a subgroup of ITT population (included all participants who received study treatment and had at least one post-baseline efficacy measurement) that included participants with MGI <=2.00 [N=39] . Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 18 | 21
Score on scale
  At week 12 with baseline MGI <=2.00 | 0.11 (0.119) | 0.21 (0.093)
  At week 24 with baseline MGI <=2.00: number analyzed (Participants) | 17 | 21
  At week 24 with baseline MGI <=2.00 | 0.10 (0.097) | 0.16 (0.082)

4. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by BI Indices in High MGI Subgroup (>2.00) at 12 and 24 Weeks
Description: as for outcome 3
Time Frame: At Week 12 and Week 24
Population: Analysis was performed on a subgroup of ITT population (included all participants who received study treatment and had at least one post-baseline efficacy measurement) that included participants with MGI >2.00 [N=52] . Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 25 | 27
Score on scale
  At week 12 with baseline MGI >2.00 | 0.11 (0.094) | 0.25 (0.144)
  At week 24 with baseline MGI >2.00 | 0.12 (0.092) | 0.21 (0.117)

5. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by Modified Gingival Index (MGI) at 12 and 24 Weeks
Description: MGI- to assess visual symptoms of gingivitis on facial and lingual surfaces of each scorable tooth (7 in each arch). 2scores recorded buccally/labially, 2scores lingually/palatally. Values presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e.,0-4). Scoring was performed using standard dental light:0=absence of inflammation,1=mild inflammation;slight change in color,little change in color; little change in texture of any portion of the marginal or papillary gingival unit,2=mild inflammation; criteria as above plus the entire marginal or papillar gingival unit,3=moderate inflammation;glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit,4=severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit,spontaneous bleeding,congestion,or ulceration. Lower scores indicate better results.
Time Frame: At Week 12 and Week 24
Population: Analysis was performed on ITT population [N=91] which included all participants who received study treatment and had at least one post-baseline efficacy measurement. Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 43 | 48
Score on scale
  At week 12 | 1.43 (0.403) | 1.87 (0.237)
  At week 24: number analyzed (Participants) | 42 | 48
  At week 24 | 1.46 (0.373) | 1.78 (0.316)

6. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by MGI Indices in Low MGI Subgroup (<=2.00) at 12 and 24 Weeks
Description: MGI-to assess gingivitis symptoms on facial, lingual surfaces of each scorable tooth(7in each arch).2 scores recorded buccally/labially(papilla,margin),2lingually/palatally(papilla,margin).Participants stratified based upon gender and baseline MGI score(Low:<=2.00,High:>2.00).Whole mouth mean of MGI calculated by-taking average overall tooth sites assessed;to compare magnitude of differences in two strata.MGI scoring:0=absence of inflammation, 1=mild inflammation;slight change in color,little change in color;little change in texture of any portion of the marginal or papillary gingival unit,2=mild inflammation;criteria as above plus the entire marginal or papillar gingival unit,3=moderate inflammation;glazing,redness,edema,and/or hypertrophy of the marginal or papillary gingival unit,4=severe inflammation;marked redness,edema and/or hypertrophy of the marginal or papillary gingival unit,spontaneous bleeding,congestion or ulceration. Lower scores indicate better results.
Time Frame: At Week 12 and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 18 | 21
Score on scale
  At week 12 with baseline MGI <=2.00 | 1.26 (0.409) | 1.74 (0.199)
  At week 24 with baseline MGI <=2.00: number analyzed (Participants) | 17 | 21
  At week 24 with baseline MGI <=2.00 | 1.29 (0.383) | 1.60 (0.319)

7. Secondary Outcome: Evaluation and Comparison of Gingival Health Measured by MGI Indices in High MGI Subgroup (>2.00) at 12 and 24 Weeks
Description: as for outcome 6
Time Frame: At Week 12 and Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 25 | 27
Score on scale
  At week 12 with baseline MGI >2.00 | 1.54 (0.364) | 1.96 (0.220)
  At week 24 with baseline MGI >2.00 | 1.57 (0.324) | 1.93 (0.231)

8. Secondary Outcome: Evaluation and Comparison of Supra-gingival Plaque Levels Measured by Overall and Inter-proximal Plaque Index (PI) at 12 and 24 Weeks
Description: Turesky Modification of Quigley Hein Plaque Index-to assess plaque on all gradable teeth. Participants rinsed the plaque in dye solution of 5milliliters(mL)of solution for 10 sec, then expectorated and rinsed with 10 mL of water for 10 sec and then expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces. Values presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e.,0-5). Disclosed plaque scored as:0=no plaque, 1=slight flecks of plaque at the cervical margin of the tooth,2=a thin continuous band of plaque (1mm or smaller) at the cervical margin of the tooth, 3=a band of plaque wider than 1mm but covering less than 1/3 of the area, 4=plaque covering at least 1/3 but less than 2/3 of the area,5=plaque covering 2/3 or more of the crown of the tooth. Lower scores indicate better results.
Time Frame: At Week 12 and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 43 | 48
Score on scale
  Overall analysis at week 12 | 2.60 (0.454) | 2.90 (0.407)
  Overall analysis at week 24: number analyzed (Participants) | 42 | 48
  Overall analysis at week 24 | 2.56 (0.527) | 2.83 (0.355)
  Interproximal analysis at week 12 | 2.82 (0.399) | 3.05 (0.354)
  Interproximal analysis at week 24 | 2.78 (0.469) | 3.00 (0.317)

9. Other Pre Specified Outcome: Number of Bleeding Sites After 12 and 24 Weeks
Description: Number of gingival bleeding sites were measured as part of bleeding index via a single examiner using a color-coded periodontal probe. The probe was engaged approximately 1 mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. For each participant, the scoring system used to measure bleeding sites is as follows: 0= no bleeding after 30 sec, 1= bleeding upon probing after 30 sec, 2= immediate bleeding observed. Lower bleeding sites indicate better results.
Time Frame: At Week 12 and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of bleeding sites
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 43 | 48
Number of bleeding sites
  At week 12 | 12.26 (10.468) | 23.92 (11.024)
  At week 24: number analyzed (Participants) | 42 | 48
  At week 24 | 12.69 (10.120) | 20.19 (9.225)

ADVERSE EVENTS:
Time Frame: From baseline up to week 24
Description: The Safety Population (N=98) included all participants who received at least 1 dose of the study product (test or reference product). Adverse Events (AEs) were regarded as treatment-emergent if they occurred on or after the first study product administration.
Arm/Group | Experimental Test Stannous Fluoride Dentifrice | Control Sodium Monofluorophosphate Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Test Stannous Fluoride Dentifrice (N=50) | Control Sodium Monofluorophosphate Dentifrice (N=48)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.